CLINICAL TRIAL: NCT02262663
Title: A Randomized, Double-blind, Parallel-group, Multi-center Study to Investigate the Pharmacodynamics, Pharmacokinetics and Safety After Daily Oral Administration of 4 Different Doses of Vilaprisan (BAY1002670) in Healthy Women of Reproductive Age
Brief Title: Study in Healthy Young Women to Investigate the Pharmacodynamics, Pharmacokinetics and Safety of Vilaprisan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 15818; 2014-000329-19 (EudraCT Number)
Record Dates: First submitted 2014-10-09; First posted 2014-10-13 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Clinical Trial, Phase I
MeSH Terms: interventions — vilaprisan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Vilaprisan [0.5mg] (Experimental): 0.5 mg BAY1002670, oral administration, one tablet to be taken daily, 84 consecutive days
  Interventions: Drug: Vilaprisan (BAY1002670)
- Vilaprisan [1mg] (Experimental): 1 mg BAY1002670, oral administration, one tablet to be taken daily, 84 consecutive days
  Interventions: Drug: Vilaprisan (BAY1002670)
- Vilaprisan [2mg] (Experimental): 2 mg BAY1002670, oral administration, one tablet to be taken daily, 84 consecutive days
  Interventions: Drug: Vilaprisan (BAY1002670)
- Vilaprisan [4mg] (Experimental): 4 mg BAY1002670, oral administration, one tablet to be taken daily, 84 consecutive days
  Interventions: Drug: Vilaprisan (BAY1002670)

INTERVENTIONS:
Drug: Vilaprisan (BAY1002670)

SUMMARY:
This is a study in healthy women of reproductive age to investigate the pharmacodynamics (mainly ovarian activity), pharmacokinetics and safety of vilaprisan after daily oral administration of 4 different doses over 84 days, using a randomized, parallel-group, multicenter design.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI): ≥ 18 and ≤ 32 kg/m² at the first screening visit
* Absence of clinically relevant abnormal findings in the pre-treatment endometrial biopsy
* Pre-treatment cycle assessed as ovulatory and not longer than 44 days

Exclusion Criteria:

* Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination or effects of the study drugs will not be normal
* Known or suspected liver disorders
* Amenorrhea for more than 3 months within the last 6 months before the first screening examination
* Clinically relevant findings (e.g. blood pressure, electrocardiogram [ECG], physical and gynecological examination, laboratory examination)
* Positive urine pregnancy test
* Regular use of medicines

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2014-10; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Hoogland score during treatment, day 9 to day 28 | Day 9 to 28
  based on maximum size of follicle-like structures, estradiol and progesterone serum concentrations
Hoogland score during treatment, day 63 to day 84 | Day 63 to 84
  based on maximum size of follicle-like structures, estradiol and progesterone serum concentrations
Hoogland score during follow up cycle 1 | 4 weeks following treatment period
  based on maximum size of follicle-like structures, estradiol and progesterone serum concentrations
Hoogland score during follow up cycle 2 | 4 weeks following follow up cycle 1
  based on maximum size of follicle-like structures, estradiol and progesterone serum concentrations
Number of subjects without bleeding/spotting | After three month treatment

SECONDARY OUTCOMES:
Exposure-response analysis of vilaprisan by population pharmacokinetic/pharmacodynamic modeling | After three month treatment
Number of subjects with TEAEs (treatment-emergent adverse events) | After three month treatment and during follow-up (up to 60 days)
Number of subjects with PAEC (progesterone-receptor-modulator associated endometrial changes) | After three month treatment and during follow-up (up to 60 days)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Berlin, State of Berlin, Germany